CLINICAL TRIAL: NCT04820374
Title: The Guiding Significance of Pupil Monitoring in the Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20210318
Record Dates: First submitted 2021-03-21; First posted 2021-03-29 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Pupil Diameter; Pupil Contraction Rate; Pupil Light Reflection
Keywords: Pupil; Cognitive Dysfunction; recovery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional extubation indications and traditional restoration indoor requirements (No Intervention)
- Extubate the tube according to the pupil index and leave the recovery room (Experimental)
  Interventions: Procedure: pupil's light and pupil diameter

INTERVENTIONS:
Procedure: pupil's light and pupil diameter — It is necessary to meet the requirement that the pupil's light reflection is slightly restored to the state of entering the room, and then the tube is extubated and the pupil diameter and the light reflection are restored to the state of entering the room, leaving the recovery room
  Arms: Extubate the tube according to the pupil index and leave the recovery room

SUMMARY:
The pupil diameter is affected by both sympathetic and parasympathetic nerves, and its latency and response amplitude mainly reflect the functional status of the parasympathetic nerve. Clinically, the diagnosis of neurological diseases can often be made based on changes in pupils.

An appropriate depth of anesthesia can cause minimal damage to the body after surgery, thereby reducing the impact on brain function and cognitive function.

The occurrence of postoperative delirium will have adverse effects on the prognosis of patients, such as prolonging the hospital stay, increasing the mortality of patients after surgery, and increasing early postoperative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients undergoing general anesthesia for tracheal intubation, aged ≥65 years, operation time ≥2 hours, ASA classification I-III, and postoperative hospital stay for at least one week.

Exclusion Criteria:

1. It is known that this study involves persons who are allergic to general anesthetics;
2. Patients with previous eye diseases;
3. Head and neck surgery is not conducive to measurement;
4. Patients with preoperative MMSE score less than 24 points or dementia due to various diseases;
5. Patients planning to undergo neurosurgery;
6. Those who use sedatives or antipsychotics before surgery;
7. Patients with known central nervous system diseases, such as mental illness; Patients with hearing or vision impairment and unable to communicate normally.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in the level of CAM-ICU scale score | 1,2,3,7 days after surgery
  First, evaluate the patient's state of consciousness based on the patient's behavior, and decide whether to proceed with the next evaluation based on the state of consciousness. If the next step is to be evaluated, ask the patient related questions to score, and evaluate whether the patient has delirium based on the score.The lower the score, the more likely the patient is to suffer from delirium.
  questions to score, and evaluate whether the patient has delirium based on the score.
  with the next evaluation based on the state of consciousness. If the next step is to be evaluated, ask the patient related questions to score, and evaluate whether the patient has delirium based on the score.
Changes in the level of Mini-Men-tal State Examination scale score | The day before surgery and 1,2,3,7 days after surgery
  Assess the cognitive function of the patient by asking questions on the patient scale.A score of 27 to 30 indicates normal cognitive function, and a score below 27 indicates cognitive dysfunction.
Changes in the level of Pittsburgh sleep quality index | The day before surgery and 1,2,3,7 days
  Assess the patient's sleep quality by asking questions on the scale.The lower the score, the more serious the sleep disorder.
Changes in the level of pupil light reflection | "before surgery", "the time of intubation", the time of extubation", "1min,3minafter intubation", "10min,20min, 30min after extubation", "the reflection of light appears""1,2,3,7 day after surgery "
Changes in the level of Polysomnography | "before surgery", "the time of intubation", the time of extubation", "1min,3min after intubation", "10min,20min, 30min after extubation", "the reflection of light appears""1,2,3,7 day after surgery "
  Through the polysomnograph, monitor the patient's sleep during anesthesia, including brain wave changes and sleep stages at different time points
Changes in the level of pupil diameter | "before surgery", "the time of intubation", the time of extubation", "1min,3minafter intubation", "10min,20min, 30min after extubation", "the reflection of light appears""1,2,3,7 day after surgery "

SECONDARY OUTCOMES:
Changes in the waveform of Narcotrend | "before surgery", "the time of intubation", the time of extubation", "1min,3min after intubation", "10min,20min, 30min after extubation", "the reflection of light appears"
  The outcome above should be measured at the time Before induction, immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
Changes in the level of Heart Rate | "before surgery", "the time of intubation", the time of extubation", "1min,3min after intubation", "10min,20min, 30min after extubation", "the reflection of light appears"
Changes in the level of Systolic Blood Pressure/Diastolic Blood Pressure(Mean Arterial Pressure) | "before surgery", "the time of intubation", the time of extubation", "1min,3min after intubation", "10min,20min, 30min after extubation", "the reflection of light appears"
Changes in the level of Oxygen saturation | "before surgery", "the time of intubation", the time of extubation", "1min,3min after intubation", "10min,20min, 30min after extubation", "the reflection of light appears"

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China